CLINICAL TRIAL: NCT06208761
Title: Effects of Triphala Supplementation and High-intensity Interval Exercise on Immune System Function and Oxidative Stress in People With Long COVID
Brief Title: Triphala Supplementation and High-intensity Interval Exercise and Immune System Function and Oxidative Stress
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Burapha University (Other)
Responsible Party: Principal Investigator, Piyapong Prasertsri, Associate Professor Dr., Burapha University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: IRB1-050/2566
Record Dates: First submitted 2023-12-21; First posted 2024-01-17 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Triphala Capsule Supplementation; High-intensity Interval Training
MeSH Terms: interventions — triphala; Dietary Supplements; High-Intensity Interval Training

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo capsule supplementation (Placebo Comparator): Participants were randomized to receive an arm. In this arm, participants consumed placebo capsule for 2 capsules daily consisting of 1 capsule (500 mg) before breakfast and 1 capsule (500 mg) before dinner, 5 days/week - separated by a couple of days, for 8 weeks. Consumption was taken at participants' dwelling.
  Interventions: Other: Triphala capsule supplementation and high-intensity interval training
- Triphala capsule supplementation (Experimental): Participants were randomized to receive an arm. In this arm, participants consumed Triphala capsule for 2 capsules daily consisting of 1 capsule (500 mg) before breakfast and 1 capsule (500 mg) before dinner, 5 days/week - separated by a couple of days, for 8 weeks. Consumption was taken at participants' dwelling.
  Interventions: Other: Triphala capsule supplementation and high-intensity interval training
- High-intensity interval training (Experimental): Participants were randomized to receive an arm. In this arm, participants received leg cycling exercise program in the form of high-intensity interval training for 28 min/day, 3 days/week for 8 weeks. Exercise training was performed at Burapha University.
  Interventions: Other: Triphala capsule supplementation and high-intensity interval training
- Triphala capsule supplementation and high-intensity interval training (Experimental): Participants were randomized to receive an arm. In this arm, participants received both Triphala capsule and high-intensity interval training in the similar extent to the Triphala capsule supplementation and high-intensity interval training arms. Consumption was taken at participants' dwelling and exercise training was performed at Burapha University.
  Interventions: Other: Triphala capsule supplementation and high-intensity interval training

INTERVENTIONS:
Other: Triphala capsule supplementation and high-intensity interval training — Triphala capsule supplementation is categorized in dietary supplement but and high-intensity interval training is included as other

SUMMARY:
One hundred and forty-one male and female participants aged 18-59 years were randomly divided into 4 groups: 1) control group: neither received exercise program nor supplement but received placebo capsule for 8 weeks 2) experiment-1: received Triphala capsule at 1,000 mg/day, before breakfast for 500 mg and before dinner for 500 mg, for consecutive 5 days/week for 8 weeks 3) experiment-2: received leg cycling exercise program in the form of high-intensity interval training (HIIT) for 28 min/day, 3 days/week for 8 weeks and 4) experiment-3: received both Triphala capsule and HIIT in the similar extent to the experiment-1 and experiment-2 groups for 8 weeks. Immune system function and oxidative stress including blood interferon-gamma (IFN-gamma), tumor necrosis factor-alpha (TNF-alpha), malondialdehyde (MDA), and protein carbonyls levels were analyzed. In addition, blood alanine aminotransferase (ALT) enzyme and creatinine levels were also analyzed for determining liver and kidney toxicity, particularly in the Triphala supplementation and combined Triphala supplementation and HIIT groups.

DETAILED DESCRIPTION:
This study aimed to investigate and compare immune system function and oxidative stress before and after supplementation with Triphala and high-intensity interval training in individuals with post COVID-19. One hundred and forty-one male and female participants aged 18-59 years were randomly divided into 4 groups: 1) control group: neither received exercise program nor supplement but received placebo capsule for 8 weeks 2) experiment-1: received Triphala capsule at 1,000 mg/day, before breakfast for 500 mg and before dinner for 500 mg, for consecutive 5 days/week for 8 weeks 3) experiment-2: received leg cycling exercise program in the form of high-intensity interval training (HIIT) for 28 min/day, 3 days/week for 8 weeks and 4) experiment-3: received both Triphala capsule and HIIT in the similar extent to the experiment-1 and experiment-2 groups for 8 weeks. Immune system function and oxidative stress including blood interferon-gamma (IFN-gamma), tumor necrosis factor-alpha (TNF-alpha), malondialdehyde (MDA), and protein carbonyls levels were analyzed. In addition, blood alanine aminotransferase (ALT) enzyme and creatinine levels were also analyzed for determining liver and kidney toxicity, particularly in the Triphala supplementation and combined Triphala supplementation and HIIT groups. Results showed that levels of IFN-gamma, TNF-alpha, MDA, and protein carbonyls before 8-week program were not different among 4 groups. After the program the levels of IFN-gamma, TNF-alpha, MDA, and protein carbonyls were significantly decreased in the Triphala supplementation, HIIT, and combined Triphala supplementation and HIIT groups (all p < 0.05). However, there were no significant differences between groups. Besides, levels of ALT enzyme and creatinine were not different among the 4 groups both before and after the 8-week program. There were also no significant differences between groups. This study concluded that in individuals with post COVID-19, Triphala supplementation at 1,000 mg/day, 5 days/week for consecutive 8 weeks can improve immune system function and alleviate oxidative stress. These outcomes are similar to those of HIIT and combined Triphala supplementation and HIIT interventions. However, prolonged investigation periods may help observing differences between interventions.

ELIGIBILITY:
Inclusion Criteria:

* Passed COVID-19 infection for at least 4 weeks with a symptom of long COVID including regular fatigue, headache, inability to concentrate, hair loss, and dyspnea (the symptom was exacerbated by exercise or concentration)
* Aged between 18 to 59 years
* Normal body mass index (BMI 18.5 to 24.9 kg/m2)

Exclusion Criteria:

* Regular exerciser (>2 times per week or >150 min per week)
* Regular intake of dietary supplements, i.e., vitamins, antioxidants, herbs
* Regular smokers or alcohol drinkers (>2 times per week)
* Food allergy, especially herbs i.e., emblic myrobalan, chebulic myrobalan, beleric myrobalan
* Hypertension, diabetes, cardiovascular disease, respiratory disease, endocrine disease, neuromuscular disease, musculoskeletal disease, liver disease, renal disease, immune disease, infectious disease, or cancer
* Current signs or symptoms of infection, i.e., fever, hyperpnea, dyspnea, and palpitations

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 141 (Actual)
Dates: Start 2023-05-09 (Actual); Primary Completion 2023-10-22 (Actual); Study Completion 2023-11-06 (Actual)

PRIMARY OUTCOMES:
Concentration of interferon-gamma | Before and after 8 weeks
  Concentration of interferon-gamma was measured in serum in pg (picogram)/mL unit
Concentration of tumor necrosis factor-alpha | Before and after 8 weeks
  Concentration of tumor necrosis factor-alpha was measured in serum in pg (picogram)/mL unit
Concentration of blood malondialdehyde | Before and after 8 weeks
  Concentration of malondialdehyde was measured in plasma in uM (micromolar) unit
Concentration of blood protein carbonyl | Before and after 8 weeks
  Concentration of protein carbonyl was measured in plasma in nmol/mg protein unit

SECONDARY OUTCOMES:
Concentration of blood alanine aminotransferase enzyme | Before and after 8 weeks
  Concentration of alanine aminotransferase enzyme was measured in serum in U/L unit
Concentration of blood creatinine | Before and after 8 weeks
  Concentration of creatinine was measured in serum in mg/dL unit

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Allied Health Sciences, Burapha University, Mueang, Changwat Chon Buri, Thailand

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers